CLINICAL TRIAL: NCT02674893
Title: Comparative Study of Gustatory Performance, Sensory Specific Satiation, Liking and Wanting in Patients With Type 2 Diabetes
Brief Title: Effect of Victoza on Dietary Preferences and Habit in Patients With Type 2 Diabetes
Acronym: GLP1 et Goût
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Exploratory protocol, convincing results, robust analysis
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Model: Parallel
Other Study IDs: BRINDISI 2013
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes; Overweight
Keywords: BMI>27; Treatment with Liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — Liraglutide; Observation

ARMS (3):
- type 2 diabetics treated with GLP1 analogue (Experimental)
  Interventions: Drug: Liraglutide
- Type 2 diabetics not treated with incretins (Active Comparator)
  Interventions: Other: Observation alone
- Healthy subjects (Other)
  Interventions: Other: Observation alone

INTERVENTIONS:
Drug: Liraglutide
  Arms: type 2 diabetics treated with GLP1 analogue
Other: Observation alone
  Arms: Healthy subjects; Type 2 diabetics not treated with incretins

SUMMARY:
This is an open-label comparative study in three parallel groups. It is expected that 90 patients and/or healthy volunteers will participate in this biomedical research.

Distribution in groups

* 30 patients with type 2 diabetes and an indication for treatment with a GLP1 analogue (group 1)
* 30 patients with type 2 diabetes (control diabetic subjects) not treated with Incretins (group 2)
* 30 healthy subjects (non-diabetics) (group 3)

This study will investigate modifications in eating behaviour induced by Liraglutide in patients who start treatment with Victoza® and certain aspects, such as liking (hedonic characteristic of a food), wanting (desire to eat a given food) and salivation in response to the presentation of a food by taking measurements at D0 (before initiation of the treatment with Liraglutide in the group concerned) then at 15 days (except for the controls), 3 months and 9 months (only for controls).

ELIGIBILITY:
Inclusion Criteria:

DIABETIC PATIENTS TREATED WITH LIRAGLUTIDE

* persons who have provided written informed consent
* aged > 18 years
* type 2 diabetes with HbA1C > 7%
* overweight (BMI > 27)
* normal renal function (creatinine clearance > 50ml/min)
* patients to be treated with Liraglutide (patients with type 2 diabetes with HbA1C > 7.5% and overweight or obesity, whose current treatment is insufficient to control the diabetes).

CONTROL DIABETIC PATIENTS

* persons who have provided written informed consent
* aged > 18 years
* type 2 diabetes with HbA1C > 7%
* overweight (BMI > 27)
* patients for whom treatment with Liraglutide is not indicated
* normal renal function (creatinine clearance > 50ml/min)

HEALTHY SUBJECTS

* persons who have provided written informed consent
* aged > 18 years

Exclusion Criteria:

DIABETIC PATIENTS TREATED WITH LIRAGLUTIDE

* type 1 diabetes
* decompensated congestive heart failure
* acute or chronic infection, progressive cancer, liver cirrhosis
* ongoing treatment with antibiotics
* smoking
* chronic alcohol abuse (>4 glasses a day)
* aversion to the products to be eaten or smelled
* poor understanding of the cognitive tasks requested
* treatment interfering with olfactogustatory performance, such as psychotropic, anti-emetic and anti-ulcer drugs
* persons without national health insurance cover
* persons under guardianship
* hypersensitivity to Liraglutide
* pregnancy, breastfeeding
* history of acute or chronic pancreatitis
* calcitonin level at selection ≥ 50 ng/L
* liver disease, defined by a level of alanine aminotransferase (ALAT) ≥ 2.5 times the upper limit of normal (ULN) for reference values

CONTROL DIABETIC PATIENTS

* type 1 diabetes,
* decompensated congestive heart failure,
* acute or chronic infection, progressive cancer, liver cirrhosis,
* ongoing treatment with antibiotics,
* smoking
* chronic alcohol abuse (> 4 glasses a day),
* aversion to the products to be eaten or smelled,
* poor understanding of the cognitive tasks requested,
* treatment interfering with olfactogustatory performance, such as psychotropic, anti-emetic and anti-ulcer drugs.
* persons without national health insurance cover
* persons under guardianship

HEALTHY SUBJECTS

* diabetes (type I and II)
* sensory disorders
* decompensated congestive heart failure,
* acute or chronic infection, progressive cancer, liver cirrhosis,
* ongoing treatment with antibiotics,
* smoking
* chronic alcohol abuse (> 4 glasses a day),
* aversion to the products to be eaten or smelled,
* poor understanding of the cognitive tasks requested,
* treatment interfering with olfactogustatory performance (psychotropic, anti-emetic, anti-ulcer drugs)
* persons without national health insurance cover
* persons under guardianship
* contra-indications to MRI, notably, but not limited to: pace maker, implantable cardiac defibrillators, neurostimulators, cochlear implants, certain implanted automated injection systems (insulin pumps), vascular intracerebral ferromagnetic clips, certain systems to regulate intravascular temperature, myopia requiring the patients to wear spectacle, history of stroke or transient ischemic attack (TIA), metallic foreign body, in particular intraocular or situated near high-risk zones (nervous system, vascular system), claustrophobia….

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Modifications in wanting | Up to 3 months

SECONDARY OUTCOMES:
Modifications in gustatory performance | Until 3 months
Modifications in liking | Until 3 months
Modifications in salivation following the presentation of foods | Until 3 months
Modifications in optimal preferences for sweet and fatty tastes | Until 3 months
Anthropometric modifications | Until 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France

REFERENCES:
- [Result] Brindisi MC, Brondel L, Meillon S, Barthet S, Grall S, Fenech C, Lienard F, Schlich P, Astruc K, Mouillot T, Jacquin-Piques A, Leloup C, Verges B, Penicaud L. Proof of concept: Effect of GLP-1 agonist on food hedonic responses and taste sensitivity in poor controlled type 2 diabetic patients. Diabetes Metab Syndr. 2019 Jul-Aug;13(4):2489-2494. doi: 10.1016/j.dsx.2019.06.021. Epub 2019 Jun 29. PMID 31405666